CLINICAL TRIAL: NCT00782990
Title: A Three Year Follow-up Prospective Open Randomized Trial of Tension-Free Vaginal Tape and Colposuspension for Primary Urodynamic Stress Incontinence
Brief Title: A 3 Year Follow-up Prospective Open Randomized Trial of TVT Versus Colposuspension for Primary Stress Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Severo Ochoa (Other)
Responsible Party: Miguel Téllez Martínez-Fornés, Hospital Severo Ochoa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVTvsBURCH_2001_HSVO
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Urinary Incontinence
Keywords: stress urinary incontinence; female incontinence; surgical treatment; Female stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

ARMS (2):
- tvt group (Active Comparator): Surgical treatment for incontinence: TVT
  Interventions: Procedure: Surgical treatment: TVT
- Burch group (Active Comparator): Surgical treatment for incontinence: Colposuspension
  Interventions: Procedure: Surgical treatment: colposuspension

INTERVENTIONS:
Procedure: Surgical treatment: TVT
  Arms: tvt group
Procedure: Surgical treatment: colposuspension
  Arms: Burch group

SUMMARY:
Objective: To compare TVT with COLPOSUSPENSION (CS) as primary treatment for stress incontinence (SUI).

Design: Randomised, open, comparative trial 3-years follow-up. Participants: 49 consecutive 35 to 70 years old women with urodynamic SUI. Setting: Urology department of a district general hospital at Leganés (Madrid), Spain.

Intervention: 24 patients randomised to TVT and 25 to CS.

DETAILED DESCRIPTION:
Background: Evidence comparing effectiveness of tension-free vaginal tape (TVT) and Burch's colposuspension (CS) in the long term follow-up is weak.

Objective: To compare TVT with CS as primary treatment for stress incontinence (SUI).

Design: Randomised, open, comparative trial 3-years follow-up. Participants: 49 consecutive 35 to 70 years old women with urodynamic SUI. Setting: Urology department of a district general hospital at Leganés (Madrid), Spain.

Intervention: 24 patients randomised to TVT and 25 to CS. Measurements: Main outcome: Assessment before treatment and at 6-months, 1-year and 3-years postoperatively with the incontinence severity symptoms index (ISS) and the incontinence impact symptoms index (IIS) Secondary outcome: 3 groups to asses cure rates: cured, improved and failure.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 35 and 70 who had completed their family with a clinical (Booney test positive) and urodynamic diagnosis of Stress Urinary Incontinence
* Previous surgery for prolapse, incontinence or bladder disease, urodynamic diagnosis of detrusor overactivity, or voiding difficulty (defined as maximum flow less than 15 ml/second or voiding pressure greater than 50 cm H2O or residual volume greater than 100 ml)
* Cystocele over grade I
* Previous hysterectomy
* Body mass index (BMI) of 40 or more
* Uncontrolled diabetes
* Neurological disease
* Recurrent urinary tract infections
* Genital atrophy precluding vaginal surgery
* Known bleeding diathesis or current anticoagulant therapy

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-01; Primary Completion 2004-10 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Subjective SUI cure evaluated with incontinence severity symptoms (ISS) and incontinence impact symptoms (IIS)

SECONDARY OUTCOMES:
Criteria were established to include patients in one of three groups: cure, improved and treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Téllez M Martínez-Fornés, urologist, Principal Investigator — Urology department. Hospital severo Ochoa.
Locations (1):
- Hospital Severo Ochoa, Leganés, Madrid, Spain